CLINICAL TRIAL: NCT06861114
Title: Exploring the Value of Urine Proteomics-based Dynamic Surveillance for Early Recurrence After Radical Surgery for Hepatocellular Carcinoma: a Prospective Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Mingxin Pan, chief physician, Zhujiang Hospital
Other Study IDs: 2025-KY-046-01
Record Dates: First submitted 2025-03-02; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: urinary proteomics; Hepatocellular carcinoma recurrence after surgery
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urinate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Urine proteomics — Patients with hepatocellular carcinoma amenable to radical resection were included according to the inclusion exclusion criteria, and preoperative urine and postoperative urine from consecutive patients were collected at the marker time (before receiving postoperative adjuvant therapy after radical surgery for hepatocellular carcinoma) and at the longitudinal time (at the time point of 3 months after radical surgery), and the different samples were preprocessed, followed by mass spectrometry-based urinary proteomics to detect the differences in urinary proteins, and the data were recorded to compare the differences.

SUMMARY:
In this study, we explored and validated the predictive value of the longitudinal monitoring model of urinary proteomics for postoperative recurrence of hepatocellular carcinoma and the predictive value of minimal residual disease (MRD) status, verified whether it is earlier than the recurrence suggested by imaging tests, and initially explored its clinical feasibility in guiding the adjuvant treatment of hepatocellular carcinoma in the postoperative period, so as to provide a new idea for the strategy of early intervention in the postoperative period of hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatocellular carcinoma whose tumor stage at the time of initial diagnosis is consistent with BCLC staging 0/stage A/stage B, who can undergo radical surgical resection, and who have not received other antitumor therapy preoperatively.

Exclusion Criteria:

* Unable to provide specimens for testing such as urine proteomics; patients with a previous diagnosis of renal or urologic disease, two or more tumors at the same time; patients with non-primary foci of liver disease. Previously received anti-tumor therapy such as targeted immunotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatocellular carcinoma whose tumor stage at the time of initial diagnosis is consistent with BCLC staging 0/stage A/stage B, who can undergo radical surgical resection, and who have not received other antitumor therapy preoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2027-12-20 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year relapse-free survival | 2-year

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No